CLINICAL TRIAL: NCT04580004
Title: The Optimization of Medications in Chronic Heart Failure Using a Website
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of personnel to run the study.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Dorsch, Assistant Professor of Clinical Pharmacy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00158766
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Optimization Group (Experimental): Patients randomized to the medication optimization group will receive an evidence-based medication recommendation intervention.
  Interventions: Other: Med Optimization Arm
- Control Group (No Intervention): Patients in the control group will receive the same intervention, delayed 2 weeks after the intervention group. During those initial 2 weeks they will act as a control.

INTERVENTIONS:
Other: Med Optimization Arm — An evidence-based medication recommendation website that is provided to the patients.
  Arms: Medication Optimization Group

SUMMARY:
Heart failure (HF) is the most common hospital discharge diagnosis among older adults in the United States. Strikingly, 2 in 5 patients are readmitted within 1-year following their first HF admission. This results in significant potentially avoidable costs to our already strained healthcare system since hospitalizations result in 70% of yearly HF management costs. One of the most common causes of readmission is lack of medication optimization. This study will determine the effectiveness of a medication optimization website.

DETAILED DESCRIPTION:
In a prospective design, 100 patients will be randomized to the intervention or usual care in a 1:1 fashion. Patients randomized to the intervention will receive an evidence-based medication recommendation intervention. Outcome measures will be collected at baseline and at 2 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction (LVEF) </= 40%

Exclusion Criteria:

* pregnancy
* active cancer with a life expectancy less than 12 months
* hospice
* chronic inotropic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
The change in medications will be measured by the Evidence Based Medicine Percent Score (EBMPS). | Change over 2 weeks
  The Evidence Based Medicine Percent Score (EBMPS) is calculated by the medications and doses the patient is taking (in points) divided by the total eligible medications based on the evidence (in points).

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Dorsch, PharmD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No